CLINICAL TRIAL: NCT05609890
Title: Effect of a Novel Formulation on Sleep Parameters Among People With Poor Sleep Quality: A Randomized Controlled Trial
Brief Title: Novel Formulation for Sleep Among People With Poor Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos O Mendivil (Other)
Collaborators: Team Foods Colombia S.A. (Industry)
Responsible Party: Sponsor-Investigator, Carlos O Mendivil, Professor of Medicine, University of Los Andes, Columbia
Organization: University of Los Andes, Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAC2422037
Record Dates: First submitted 2022-08-25; First posted 2022-11-08 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Sleep; Sleep Disorder; Insomnia; Quality of Life; Poor Quality Sleep
Keywords: Sleep; Supplement; Nutraceutical; Health; Quality of life; Actigraphy
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Masking Description: The participants and the investigator who will provide the intervention and collect the data will be masked about interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): A formulation made of natural components. Each sachet contains saffron, tea extract, lemon balm and valerian.
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): Placebo sachet will contain inert excipient.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Supplement: a mixture of saffron, tea extract, lemon balm and valerian.
  Dose: The participant will take one sachet every day, one hour before going to bed, for six weeks.
  Arms: Active intervention
Other: Placebo — Placebo sachet
  Dose: The participant will take one sachet everyday, one hour before going to bed, for six weeks.
  Arms: Placebo

SUMMARY:
Sleep disorders are highly prevalent all around the world and have a strong negative impact on quality of life (QoL). In Colombia, up to 60% of adults report any sleep disturbance and more than 45% have required medical assistance for this. There is abundant anecdotal and scientific evidence supporting the efficacy and safety of several plant extracts on sleep quality. In this context, the development of safe and effective natural products may have a positive impact on sleep and general QoL.

DETAILED DESCRIPTION:
It is estimated that up to 90% of people will have a sleep concern over their adult life. According to a worldwide survey, one out of two people report unsatisfactory sleep. In Colombia, a Latin American country, more than 60% of adults report sleep concerns. For a long time, positive effects on sleep of plant extracts have been described, and more recently their mechanisms of action and safety have been largely elucidated. This study aims to assess the efficacy and safety of a supplement formulation based on natural products (Saffron, Tea extract, Lemon Balm and Valerian) on objective and subjective sleep parameters.

This is a randomized, doble-blind, placebo controlled clinical trial. The primary outcome is sleep efficiency. A sample size of 60 participants is needed for having a power of 95%, a one type error of 5% and a minimal difference of at least 2.8% between groups in the primary outcome. As we estimate a loss to follow-up of 10%, 66 participants will be enrolled. The main inclusion criteria will be having a poor sleep quality demonstrated as having a Pittsburgh Sleep Quality Index (PSQI) equal to or greater than five. In a random allocation design, one group of participants will receive the active intervention and the other one will receive a placebo with similar organoleptic features. The study will be executed in three main phases: First, a run-in phase where eligible participants will receive the active intervention during one week, and only those with adherence 85% or greater continue to the next phase. Second, a wash-out phase in which participants will not receive any intervention but actigraphic data will be collected. Finally, in the third (intervention) phase participants will be randomized following a minimization algorithm to the active or placebo group, to be taken for six weeks. Subjective and objective sleep variables will be measured at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18, male or female.
* PSQI >=5
* Provision of informed consent
* Adherence >= 85%

Exclusion Criteria:

* Medical history of a specific sleep disorder according to the DSM-5
* Taking any specific pharmacologic treatment to improve sleep or planning to take it in the next two months
* Medical history of generalized anxiety disorder, depression or other serious psychiatric / neurological disease
* Uncontrolled hypothyroidism
* Medical history of deficit or excess of corticosteroids (Cushing syndrome, Addison syndrome, chronic steroid use)
* Alcohol intake (more than two standard drinks/day, on average)
* Caffeine intake more than 400 mg per day, on average
* Frequent sleep deprivation over the last two months
* Women with desire to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Baseline (week 0) - Final (week 6)
  The change (Week 6 - baseline) in Sleep Efficiency (the ratio of total sleep time to time in bed)

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) (0-21) higher scores means worse sleep quality | Baseline (week 0) - Final (week 6)
  Change from baseline in the PSQI
Short Form-36 Quality of Life score (SF-36) (0-100), higher score means better quality of life | Baseline (week 0) - Final (week 6)
  Change in QoL measured by the 36-Item Short Form Survey (SF-36)
Morning salivary cortisol | Baseline (week 0) - Final (week 6)
  Change in salivary cortisol (as a measurement of response to stress)
Blood creatinine | Baseline (week 0) - Final (week 6)
  Change in blood creatinine
Blood alanine amino transferase | Baseline (week 0) - Final (week 6)
  Change in blood alanine amino transferase

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, School of Medicine, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz AJ, Sepulveda MA, Martinez PH, Munoz MC, Mendoza LO, Centanaro OP, Carrasco LF, Garcia JC. Prevalence of sleep complaints in Colombia at different altitudes. Sleep Sci. 2016 Apr-Jun;9(2):100-5. doi: 10.1016/j.slsci.2016.05.008. Epub 2016 Jun 4. PMID 27656274
- [Background] Ong JL, Lau T, Massar SAA, Chong ZT, Ng BKL, Koek D, Zhao W, Yeo BTT, Cheong K, Chee MWL. COVID-19-related mobility reduction: heterogenous effects on sleep and physical activity rhythms. Sleep. 2021 Feb 12;44(2):zsaa179. doi: 10.1093/sleep/zsaa179. PMID 32918076
- [Background] Medic G, Wille M, Hemels ME. Short- and long-term health consequences of sleep disruption. Nat Sci Sleep. 2017 May 19;9:151-161. doi: 10.2147/NSS.S134864. eCollection 2017. PMID 28579842
- [Background] Meerlo P, Sgoifo A, Suchecki D. Restricted and disrupted sleep: effects on autonomic function, neuroendocrine stress systems and stress responsivity. Sleep Med Rev. 2008 Jun;12(3):197-210. doi: 10.1016/j.smrv.2007.07.007. Epub 2008 Jan 25. PMID 18222099
- [Background] McCoy JG, Strecker RE. The cognitive cost of sleep lost. Neurobiol Learn Mem. 2011 Nov;96(4):564-82. doi: 10.1016/j.nlm.2011.07.004. Epub 2011 Aug 22. PMID 21875679
- [Background] Meng L, Zheng Y, Hui R. The relationship of sleep duration and insomnia to risk of hypertension incidence: a meta-analysis of prospective cohort studies. Hypertens Res. 2013 Nov;36(11):985-95. doi: 10.1038/hr.2013.70. Epub 2013 Sep 5. PMID 24005775
- [Background] Pan XL, Nie L, Zhao SY, Zhang XB, Zhang S, Su ZF. The Association Between Insomnia and Atherosclerosis: A Brief Report. Nat Sci Sleep. 2022 Mar 15;14:443-448. doi: 10.2147/NSS.S336318. eCollection 2022. PMID 35313542
- [Background] Hargens TA, Kaleth AS, Edwards ES, Butner KL. Association between sleep disorders, obesity, and exercise: a review. Nat Sci Sleep. 2013 Mar 1;5:27-35. doi: 10.2147/NSS.S34838. Print 2013. PMID 23620691
- [Background] Knutson KL. Does inadequate sleep play a role in vulnerability to obesity? Am J Hum Biol. 2012 May-Jun;24(3):361-71. doi: 10.1002/ajhb.22219. Epub 2012 Jan 24. PMID 22275135
- [Background] Schipper SBJ, Van Veen MM, Elders PJM, van Straten A, Van Der Werf YD, Knutson KL, Rutters F. Sleep disorders in people with type 2 diabetes and associated health outcomes: a review of the literature. Diabetologia. 2021 Nov;64(11):2367-2377. doi: 10.1007/s00125-021-05541-0. Epub 2021 Aug 16. PMID 34401953
- [Background] Lin CL, Chien WC, Chung CH, Wu FL. Risk of type 2 diabetes in patients with insomnia: A population-based historical cohort study. Diabetes Metab Res Rev. 2018 Jan;34(1). doi: 10.1002/dmrr.2930. Epub 2017 Oct 4. PMID 28834008
- [Background] Aggarwal S, Loomba RS, Arora RR, Molnar J. Associations between sleep duration and prevalence of cardiovascular events. Clin Cardiol. 2013 Nov;36(11):671-6. doi: 10.1002/clc.22160. Epub 2013 Oct 1. PMID 24122853
- [Background] Choi Y, Choi JW. Association of sleep disturbance with risk of cardiovascular disease and all-cause mortality in patients with new-onset type 2 diabetes: data from the Korean NHIS-HEALS. Cardiovasc Diabetol. 2020 May 13;19(1):61. doi: 10.1186/s12933-020-01032-5. PMID 32404104
- [Background] Mogavero MP, DelRosso LM, Fanfulla F, Bruni O, Ferri R. Sleep disorders and cancer: State of the art and future perspectives. Sleep Med Rev. 2021 Apr;56:101409. doi: 10.1016/j.smrv.2020.101409. Epub 2020 Nov 28. PMID 33333427
- [Background] Rod NH, Vahtera J, Westerlund H, Kivimaki M, Zins M, Goldberg M, Lange T. Sleep disturbances and cause-specific mortality: Results from the GAZEL cohort study. Am J Epidemiol. 2011 Feb 1;173(3):300-9. doi: 10.1093/aje/kwq371. Epub 2010 Dec 30. PMID 21193534
- [Background] Chattu VK, Manzar MD, Kumary S, Burman D, Spence DW, Pandi-Perumal SR. The Global Problem of Insufficient Sleep and Its Serious Public Health Implications. Healthcare (Basel). 2018 Dec 20;7(1):1. doi: 10.3390/healthcare7010001. PMID 30577441
- See also: Filip I, Tidman M, Saheba N, Bennet H, Wick B, Rouse N, Patriche D, Radfar A. Public health burden of sleep disorders underreported problem. J Public Health 2016;25:243-248. — https://www.infona.pl/resource/bwmeta1.element.springer-doi-10_1007-S10389-016-0781-0
- See also: Koninklijke Philips N.V. Wake up call: global sleep satisfaction trends. Philips Global Survey [Internet] 2020 [consultado 2022 junio 28]. — https://www.philips.com/c-dam/b2c/master/experience/smartsleep/world-sleep-day/2020/2020-world-sleep-day-report.pdf